CLINICAL TRIAL: NCT04733729
Title: Epidemiology of COVID-19 Infection in Patients With Hematological Malignancies: A European Haematology Association Survey
Brief Title: Covid-19 in Hematological Malignancies
Acronym: EPICOVIDEHA
Status: Recruiting | Type: Observational
Sponsor: Sorveglianza Epidemiologica Infezioni Fungine Emopatie Maligne (Other)
Collaborators: European Hematology Association (Unknown)
Responsible Party: Principal Investigator, LIVIO PAGANO, Associated Professor of Hematology, Catholic University of the Sacred Heart
Other Study IDs: EHA-IDWG
Record Dates: First submitted 2021-01-31; First posted 2021-02-02 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: COVID-19 Infection in Hematological Malignancies Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The overall purpose of this project is to better understand the epidemiology of COVID-19 in patients with hematological malignancies (including hematopoietic stem cell transplant recipients) in the different European Countries. The results obtained will allow us to better know the prevalence of this complication in the different categories of patients with hematological malignancies (HMs). In order to attain the objectives previously described we will develop a multicentre, international, observational, retrospective and prospective study of consecutive cases of COVID-19 among HMs. There will be a clinical follow-up of the patients included in this study to observe the survival rate. Data collected form this study will be evaluated with a descriptive analysis.

DETAILED DESCRIPTION:
At the moment, few data on the epidemiology of SARS-CoV-2 infection in patients suffering from hematological malignancies are available. However, the COVID-19 pandemic presents unique challenges and opportunities on hematological malignancies. The future trajectory of this pandemic appears to be growing and hematology communities must continue to prepare for its spread In this project, we will implement cooperation between all members of the hematology departments both within the EHA and outside it, in order to evaluate the epidemiological data on the incidence and outcome in patients with hematological malignancies infected with SARS-CoV-2.

We will provide useful information to inform the individualized plan for patients with hematological malignancies.

We aim to evaluate the epidemiology and outcomes of patients with HM infected with COVID-19,estimate the incidence and type of disease, assess the acute and long-term mortality rate and estimate the overall mortality rate of cases.

This is a cohort retrospective/prospective survey. In the retrospective phase of the study, participating centers will retrospectively review episodes of COVID-19 disease that occurred in patients with hematological malignancies identified at their institutions from February 2020 to December 2020. In the prospective phase of the study, the researchers will include episodes of COVID-19 disease from the start of the study through December 31, 2021.

The study population will need to be over 18 with hematological malignancies and SARS-CoV-2 An electronic database with anonymization will be created and available to collect all information with single access for each participating institution. The data collected will be demographic data,epidemiological factors, admission information, COVID-19 disease severity, history of hematological malignancies, disease status with past / current treatments, and 30 days of diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years of age.
* History of hematological malignancies (acute leukemias, myelodysplastic syndromes, myeloproliferative neoplasms, lymphomas, myeloma, chronic myeloprolipherative disorders) at any stage/status.
* Active hematological malignancies at any stage/status.
* Diagnosis of hematological malignancy (acute leukemias, myelodysplastic syndromes, myeloproliferative neoplasms, lymphomas, myeloma, chronic myeloprolipherative disorders) at any stage/status.
* SARS-CoV-2 positive test (nasopharyngeal, BAL, fecal), documented by Real-Time Reverse Transcriptase (RT)-PCR Diagnostic Panels.

Exclusion Criteria:

* Hematological diseases, other than hematological malignancies.
* Not tested positive for SARS-CoV-2
* Patients "off therapy" for more than 5 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: No formal sample size is planned for this study because not only the main hypothesis will be assessed. However, this is a multicentre cohort study on a high incident disease, with an elevated expected number of events (death, complications, and co-infections) to be observed. So more than 2000 patients are expected to be included.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Epidemiology of COVID-19 infection in patients with hematological malignancies | 2020 (1 year)
  to evaluate the epidemiology of COVID infection among all hema malignancies patients subgroups

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - ASST-Spedali Civili, Brescia
  - AOU Policlinico Federico II, Napoli
  - Fondazione Policlinico A. Gemelli IRCCS, Rome
  - Istituto Nazionale Tumori Regina Elena IFO, Rome
  - Osp. di Circolo-Fondazione Macchi, Varese
  - AOUI Verona, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Passamonti F, Cattaneo C, Arcaini L, Bruna R, Cavo M, Merli F, Angelucci E, Krampera M, Cairoli R, Della Porta MG, Fracchiolla N, Ladetto M, Gambacorti Passerini C, Salvini M, Marchetti M, Lemoli R, Molteni A, Busca A, Cuneo A, Romano A, Giuliani N, Galimberti S, Corso A, Morotti A, Falini B, Billio A, Gherlinzoni F, Visani G, Tisi MC, Tafuri A, Tosi P, Lanza F, Massaia M, Turrini M, Ferrara F, Gurrieri C, Vallisa D, Martelli M, Derenzini E, Guarini A, Conconi A, Cuccaro A, Cudillo L, Russo D, Ciambelli F, Scattolin AM, Luppi M, Selleri C, Ortu La Barbera E, Ferrandina C, Di Renzo N, Olivieri A, Bocchia M, Gentile M, Marchesi F, Musto P, Federici AB, Candoni A, Venditti A, Fava C, Pinto A, Galieni P, Rigacci L, Armiento D, Pane F, Oberti M, Zappasodi P, Visco C, Franchi M, Grossi PA, Bertu L, Corrao G, Pagano L, Corradini P; ITA-HEMA-COV Investigators. Clinical characteristics and risk factors associated with COVID-19 severity in patients with haematological malignancies in Italy: a retrospective, multicentre, cohort study. Lancet Haematol. 2020 Oct;7(10):e737-e745. doi: 10.1016/S2352-3026(20)30251-9. Epub 2020 Aug 13. PMID 32798473
- [Background] Garcia-Suarez J, de la Cruz J, Cedillo A, Llamas P, Duarte R, Jimenez-Yuste V, Hernandez-Rivas JA, Gil-Manso R, Kwon M, Sanchez-Godoy P, Martinez-Barranco P, Colas-Lahuerta B, Herrera P, Benito-Parra L, Alegre A, Velasco A, Matilla A, Alaez-Uson MC, Martos-Martinez R, Martinez-Chamorro C, Susana-Quiroz K, Del Campo JF, de la Fuente A, Herraez R, Pascual A, Gomez E, Perez-Oteyza J, Ruiz E, Alonso A, Gonzalez-Medina J, Martin-Buitrago LN, Canales M, Gonzalez-Gascon I, Vicente-Ayuso MC, Valenciano S, Roa MG, Monteliu PE, Lopez-Jimenez J, Escobar CE, Ortiz-Martin J, Diez-Martin JL, Martinez-Lopez J; Asociacion Madrilena de Hematologia y Hemoterapia (AMHH). Impact of hematologic malignancy and type of cancer therapy on COVID-19 severity and mortality: lessons from a large population-based registry study. J Hematol Oncol. 2020 Oct 8;13(1):133. doi: 10.1186/s13045-020-00970-7. PMID 33032660
- [Background] Kuderer NM, Choueiri TK, Shah DP, Shyr Y, Rubinstein SM, Rivera DR, Shete S, Hsu CY, Desai A, de Lima Lopes G Jr, Grivas P, Painter CA, Peters S, Thompson MA, Bakouny Z, Batist G, Bekaii-Saab T, Bilen MA, Bouganim N, Larroya MB, Castellano D, Del Prete SA, Doroshow DB, Egan PC, Elkrief A, Farmakiotis D, Flora D, Galsky MD, Glover MJ, Griffiths EA, Gulati AP, Gupta S, Hafez N, Halfdanarson TR, Hawley JE, Hsu E, Kasi A, Khaki AR, Lemmon CA, Lewis C, Logan B, Masters T, McKay RR, Mesa RA, Morgans AK, Mulcahy MF, Panagiotou OA, Peddi P, Pennell NA, Reynolds K, Rosen LR, Rosovsky R, Salazar M, Schmidt A, Shah SA, Shaya JA, Steinharter J, Stockerl-Goldstein KE, Subbiah S, Vinh DC, Wehbe FH, Weissmann LB, Wu JT, Wulff-Burchfield E, Xie Z, Yeh A, Yu PP, Zhou AY, Zubiri L, Mishra S, Lyman GH, Rini BI, Warner JL; COVID-19 and Cancer Consortium. Clinical impact of COVID-19 on patients with cancer (CCC19): a cohort study. Lancet. 2020 Jun 20;395(10241):1907-1918. doi: 10.1016/S0140-6736(20)31187-9. Epub 2020 May 28. PMID 32473681
- [Derived] van Doesum JA, Salmanton-Garcia J, Marchesi F, Di Blasi R, Falces-Romero I, Cabirta A, Farina F, Besson C, Weinbergerova B, Van Praet J, Schonlein M, Lopez-Garcia A, Lamure S, Guidetti A, De Ramon-Sanchez C, Batinic J, Gavriilaki E, Tragiannidis A, Tisi MC, Plantefeve G, Petzer V, Ormazabal-Velez I, Marques de Almeida J, Marchetti M, Maertens J, Machado M, Kulasekararaj A, Hernandez-Rivas JA, Gomes da Silva M, Fernandez N, Espigado I, Drgona L, Dragonetti G, Metafuni E, Calbacho M, Blennow O, Wolf D, van Anrooij B, Nunes Rodrigues R, Nordlander A, Martin-Gonzalez JA, Lievin R, Jimenez M, Grafe SK, Garcia-Sanz R, Cordoba R, Rahimli L, van Meerten T, Cornely OA, Pagano L. Impact of SARS-CoV-2 vaccination and monoclonal antibodies on outcome post-CD19-directed CAR T-cell therapy: an EPICOVIDEHA survey. Blood Adv. 2023 Jun 13;7(11):2645-2655. doi: 10.1182/bloodadvances.2022009578. PMID 37058479
- See also: COVID-19 in pediatric malignancies — https://global.stjude.org/en-us/global-covid-19-observatory-and-resource-center-for-childhood-cancer/registry.html
- See also: ASH webpage on COVID in hematology — https://www.hematology.org/covid-19/ash-astct-covid-19-and-vaccines